CLINICAL TRIAL: NCT03561376
Title: Zinc Oxide Versus Petrolatum Following Skin Surgery: A Head-to-head, Prospective, Split-scar Study
Brief Title: Zinc Oxide Versus Petrolatum Following Skin Surgery
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Melissa Pugliano-Mauro (Other)
Responsible Party: Sponsor-Investigator, Melissa Pugliano-Mauro, Assistant Professor, Director, Mohs Surgery Program, Director Mohs Micrographic Surgery and Dermatologic Oncology Fellowship, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19050135
Record Dates: First submitted 2018-05-07; First posted 2018-06-19 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Surgical Incision; Surgery--Complications; Surgical Wound; Surgical Site Infection; Scar; Hypertrophic Scar
Keywords: Scar
MeSH Terms: conditions — Surgical Wound; Surgical Wound Infection; Cicatrix; Cicatrix, Hypertrophic

STUDY DESIGN:
Intervention Model Description: Split scar study (petrolatum vs. zinc oxide)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm - split scar study (Other): Surgical closures, at least 4.5cm in length, will be split and zinc oxide ointment applied to half and petrolatum ointment to the other half
  Interventions: Drug: Topical zinc oxide vs. petrolatum post-surgical scars

INTERVENTIONS:
Drug: Topical zinc oxide vs. petrolatum post-surgical scars — Following linear closure on non-scalp skin with scar length > 4.5 cm, incision site will be "split" and petrolatum applied to one half and zinc oxide ointment to the other half daily for one month following surgery.

SUMMARY:
Patients undergoing routine surgery in the Department of Dermatology for any indication on non-scalp skin and closed in linear fashion with scar greater than or equal to 4.5cm in length will be invited to participate in this split scar, head to head study comparing zinc oxide and petrolatum. Patients will apply respective ointments to each half of scar daily for one month and maintain a log of these activities. They will be seen at 1 week, 4 weeks, 8 weeks, and 6 months post-operatively for photographic scar assessment and to complete the patient portion of the Patient and Observer Scar Assessment Scale (POSAS), a quantitative objective assessment of scar appearance. Trained observers (board-certified dermatologists) will score the observer portion of the scale. POSAS outcomes, post-operative infections, linear density of epidermal seal will be assessed at the 1 week, 4 weeks, 8 weeks, and 6 months post-operative periods and compared between the two groups. Participants will have parking validated for all visits and upon completion of all portions of the study will receive a standardized skin care gift bag containing samples for hypoallergenic skin care products (washes, moisturizers, etc.).

DETAILED DESCRIPTION:
Patients who have undergone dermatologic excision for any indication with or without Mohs micrographic surgical technique and surgically closed in linear fashion with scar length of greater than or equal to 4.5cm on any site but the scalp will be approached for enrollment in the study. Any closure in which one half of the linear scar appears grossly unequal to or worse than the other (due to any number of causes, such as suture technique, etc.) will be excluded from the study. Any patient whose surgical procedure was deemed as having high risk of post-surgical infection would also be excluded from the study as well as those with known history of topical zinc allergy. Consent will be obtained with one of the trained co-investigators. Included in this consent will be consent to collection of basic patient medical data pertinent to wound healing/scar formation will be obtained, such as history of keloids, smoking, history of diabetes mellitus, history of cancer and/or on chemotherapy, history of transplant, and immunosuppressive status, etc. for the purposes of this research. Risk to patients using zinc oxide ointment has been deemed by the FDA as minimal. Of note, zinc oxide ointment currently is the gold standard treatment for erosive diaper dermatitis on newborns and infants. It is generally deemed safe clinically and its application to other clinical settings outside of diaper rash has not been explored.

Upon providing consent for the study, the patient's surgical closure will be demarcated with sterile inked pen and "V" will be drawn on one end and "Z" on the other. The control, standard of care petrolatum (i.e. Vaseline) will be applied to the side indicated by "V" and the experimental treatment zinc oxide will be applied to the "Z" side. As a general rule, if oriented longitudinally, "Z" will mark distal, "V" will mark proximal. If oriented horizontally (left to right), "V" will mark the left side, "Z" the right. The ointments and standard pressure dressing will be administered in clinic upon closure and consent/enrollment. Patients will be sent home with package containing standard wound dressing materials as well as both zinc oxide and petrolatum.

Patients will be sent home with instructions and wound care materials to perform the following: (1) Keep post surgical pressure dressing in place for 48 hours (2) Gentle soap and water cleansing after 48 hours once daily (3) With daily dressing changes self apply zinc oxide ointment to side indicated by "Z" and petrolatum (vaseline) to side indicated by "V" (3b) Patient will be encouraged to re-mark site Z and V to serve as reminder to enhance compliance (4) Patient will sign off on daily log twice: once upon application of zinc oxide to Z side and upon application of petrolatum to V side. (5) Patient will perform daily dressing changes as above for one month. The application of daily ointment with or without dressing is also routine standard of care at the present time. Draft of patient instructions has been included with this submission.

Patients will be seen at the routine standard of care visit 7 days post-op for suture removal. At this point in time, accompanying dressing will be taken down, cleansed with sterile saline, and patient wounds will be photographed under standardized conditions, with avoidance of any clue as to which ointment was applied to which side. In addition, patients will perform the patient portion of the POSAS (Patient and Observer Scar Assessment Scale v2.0, a validated measure of scar cosmesis, with 6 to 60 scale, with low numbers represent that scar appears most similar to normal skin, whereas 60 indicates that the scar is visually furthest from normal skin, i.e. worst possible scar). Patients will also follow-up at 4 weeks, 8 weeks, and 6 months post-operatively for scar assessment. Patient parking will be validated. For patients requesting optimal close clinical follow-up for post-surgical scars, this appointment schedule represents the highest standard of care. At these visits, photographs will be obtained, and patients will again be asked to complete the patient portion of the POSAS scale. Upon completion of the six month follow-up visit for this pilot study, patients will be given a basic skin care product sample gift bag, containing a standardized collection of samples of hypoallergenic washes and moisturizers. Of note, if a patient is unable to return for the final six month follow-up visit, patients will be allowed to submit electronic photographs (non-standardized, self taken) with clear instructions to send via secure message via MyUPMC, a secure interface allowing for communication between patient's and doctors within the UPMC (University of Pittsburgh Medical Center) network. This option is to be reserved as a last resort. Patients will not receive the gift bag if unable to return for this final study visit. Please note that patient obtained and entered photographs are routinely used clinically for remote assessment of skin disorders for routine clinical follow-up.

Board-certified dermatologists at the end of the study will evaluate the photographs obtained at a later point in the study. Through photographic and/or edited technique if necessary, they will be blinded to which side received zinc oxide and which side received petrolatum. Indeed, the POSAS has been validated with photographic use. In addition, an estimation of the linear proportion of epidermal seal will be evaluated visually based on clinical exam and/or photographs. Specifically, the length of the wound will be measured at this visit and distance of scar containing non grossly apposed skin edges will be measured. The sum of length of non-sealed areas within the V side and within the Z side will be calculated. In addition, clinical evidence of surgical site infection, wound disruption, and/or any other post-surgical complications will be documented.

Upon completion of study visits, POSAS score, epidermal seal, and other clinical data will be statistically analyzed. Compliance rates will be calculated. Primary outcome of POSAS vs. % epidermal seal will be utilized. A total of 30 participants has been established as a goal for this pilot study with guidance from the Clinical and Translational Science Institute at the University of Pittsburgh Medical Center.

The standardized post surgical scar assessment tool (SCAR, Scar Cosmesis Assessment and Rating) will be utilized to objectively record scar outcomes. In addition, photographs of the surgical sites will be taken at each visit. In exchange for their participation, all patient wound care materials will be provided by the clinic.

These research procedures will take place in the surgical suites of the UPMC Falk Dermatology Office Building and the UPMC St. Margaret's Dermatology Office Building. These activities are to take place during the 2018-19 academic year.

Clinical staff at both sites will be involved in the conduct of the study. Patients referred/scheduled to see faculty dermatologic surgeon Dr. Melissa Pugliano-Mauro will be the population pool.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Linear closure, non-scalp site
3. ≥ 4.5 cm in length (final incision/closure length)
4. End to end symmetry (surgical site is not grossly asymmetric from end to end)
5. Grossly uninfected site

Exclusion Criteria:

1. ≤ 18 years
2. Visibly asymmetric linear scar
3. Grossly infected surgical site
4. History of allergy to topical zinc oxide

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
POSAS (patient and observer scar assessment score) | 8 weeks
  Patient and observer scar assessment score. Range from 6-60. Higher score indicates greater patient satisfaction and better overall cosmesis of scar. Please note there is an observer and patient POSAS score. Both range from 6-60. The observer scale grades the apparent vascularity, pigmentation, thickness, relief, pliability, and surface area of the scar. The patient scale evaluate the patient's perception of pain, itching, color, stiffness, thickness, irregularity associated with the scar. Each item is graded from 1-10 for a combined minimum to maximum of 6-60.
Percentage of epidermal linear seal | 1 week
  % of linear scar that has fully sealed across surgical defect based on visual inspection. 0-100%. Higher percentage reflects greater proportion of visually sealed epidermis upon surgical closure.
POSAS (patient and observer scar assessment score) change between 8 weeks and six months | To be assessed at 8 weeks and six months post-operative follow-up
  Will assess for change in POSAS between weeks 8 and six months follow-up. The score will range from 0-54
Change in % epidermal linear seal between weeks 1 and 4 post-operative | weeks 1 and 4 weeks post-operative
  Will assess change in % linear epidermal seal between weeks 1 and 4. The score will range from 0-100%.
POSAS (patient and observer scar assessment score) | Six months post-operative follow-up
  Range from 6-60. Higher score indicates greater patient satisfaction and better overall cosmesis of scar
Percentage of epidermal linear seal | 4 weeks
  % of linear scar that has fully sealed across surgical defect based on visual inspection. 0-100%. Higher percentage reflects greater proportion of visually sealed epidermis upon surgical closure.

SECONDARY OUTCOMES:
Surgical site infection | 1 week, 4 weeks, 8 weeks, six months post-operatively
  As above. Any erythema, pus formation, or skin changes necessitating topical or systemic antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Crow, MD, Principal Investigator — Resident Physician, PGY-3
Locations (1):
- UPMC Dermatology St. Margaret, Pittsburgh, PA, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kantor J. The SCAR (Scar Cosmesis Assessment and Rating) scale: development and validation of a new outcome measure for postoperative scar assessment. Br J Dermatol. 2016 Dec;175(6):1394-1396. doi: 10.1111/bjd.14812. Epub 2016 Oct 17. No abstract available. PMID 27292082
- [Background] Thompson CB, Wiemken TL, Brown TS. Effect of Postoperative Dressing on Excisions Performed on the Leg: A Comparison Between Zinc Oxide Compression Dressings Versus Standard Wound Care. Dermatol Surg. 2017 Nov;43(11):1379-1384. doi: 10.1097/DSS.0000000000001209. PMID 28654576